CLINICAL TRIAL: NCT03821207
Title: The Effect of Abdominal Massage and Exercise on Primary Dysmenorrhea in University Students: A Randomised Controlled Study
Brief Title: The Effect of Abdominal Massage and Exercise on Primary Dysmenorrhea in University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Meryem Kurek eken, Associated Proffesor, Aydin Adnan Menderes University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2018/1357
Record Dates: First submitted 2018-12-30; First posted 2019-01-29 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Primary Dysmenorrhea
Keywords: Abdominal massage; Exercise; Primary Dysmenorrhea
MeSH Terms: conditions — Motor Activity | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Randomised Controlled Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The exercise group (Active Comparator): The group will be instructed to perform stretching exercises including the pelvic and lumbar regions 3 times a day for the first 3 days of the menstrual cycle
  Interventions: Behavioral: The exercise group
- The abdominal massage group (Active Comparator): The group will be instructed to massage the abdomen for 10 mins a day on the first 3 days of the menstrual cycle.The massage is to be applied as effleurage (light touch) clockwise over the abdomen
  Interventions: Behavioral: The abdominal massage group
- The control group (Placebo Comparator): The control group will perform no exercise or massage.
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: The exercise group — The students will make exercise during the first three days of the menstrual period
  Arms: The exercise group
Behavioral: The abdominal massage group — The students will make abdominal massage during the first three days of the menstrual period
  Arms: The abdominal massage group
Behavioral: Control Group — The students will nor massage or exercise
  Arms: The control group

SUMMARY:
The study will planing to determine the advantages of abdominal massage and exercise on primary dysmenorrhea in university students, and to evaluate whether one of these applications is superior to the other.

DETAILED DESCRIPTION:
The students included in the study will be randomly separated into 3 groups using a computer-based randomisation plan (www.randomization.com).

Those included in the massage group will be instructed to massage the abdomen for 10 mins a day on the first 3 days of the menstrual cycle. The massage is to be applied as effleurage (light touch) clockwise over the abdomen from over the abdominal wall to the intestinal area.

The students in the exercise group will be instructed to perform stretching exercises including the pelvic and lumbar regions 3 times a day for the first 3 days of the menstrual cycle.

The control group will perform no exercise or massage. The applications will be demonstrated to the participants by a physiotherapist. Throughout the study period, the students will be followed up to ensure that the applications are being made. Follow-up of the applications of abdominal massage and stretching exercises applied by there searcher physiotherapist according to the study plan will be conducted by the researchers.

The participants will be informed how to apply the massage and perform the exercises and that these applications will cause no side-effects. They will also be informed that participation in the study is voluntary and they can withdraw from the study at any time.

The study will include volunteer female students, aged 18- 20 years, with regular menstrual cycles, who record ≥ 6 points on VAS in the first 3 days of at least 2 of the last 3 menstrual cycles and will not use analgesics during the study.

Data Collection Tools Personal Information Form: This form was prepared by the researchers in accordance with previous reports in literature to include 5 socio-demographic items and 14 items related to the menstrual history (age of menarche, frequency of painful menstruation, amount of bleeding, family history of painful menstruation, methods of dealing with the pain, etc).

Visual Analog Scale (VAS):This scale is a simple method used in the measurement of pain severity and in the follow-up of pain. The patient is instructed to mark the severity of pain on a 10cm horizontal line, where 0= non pain and 10= intolerable pain.

Dysmenorrhea Symptom List:This list was prepared by the researchers in accordance with literature to evaluate the efficacy of the application and includes the findings seen in the presence of dysmenorrhea in females. Each finding is scored from 0-3 as 0= non symptom, 1= mild symptom that does not affect daily activity, 2 = mild non-debilitating symptom that affects daily activity, 3= totally debilitating severe symptom.

Amount of Menstrual Blood: As it is impossible to measure blood lost during menstruation in a laboratory environment, a pictorial blood loss evaluation table will be used,which is a practical and low-cost method with a high accuracy rate. The pictorial blood loss evaluation table was developed to show the degree of soiling. The participants will be given detailed instructions of how to use these forms and will be checked as to whether or not they have understood by being instructed to record a bleeding pattern described by the researchers (eg, mark on the table that in the first 2 days you have used 5 pads completely soiled and in the following 3 days, 2 half pads and 1 with staining). The pictorial index score is calculated by giving points of 1, 5 and 20 to mild, moderately and heavily soiled pads respectively, and scores of 1 and 5 for small and large clots. A cut-off value of 100 will be used. To reduce misinterpretations resulting from the use of different pads, all the participants will be recommended to use the same brand of sanitary pad.

ELIGIBILITY:
Inclusion Criteria:

Regular menstrual cycles Record ≥ 6 points on VAS in the first 3 days of at least 2 of the last 3 menstrual cycles Not use analgesics during the study period

Exclusion Criteria:

Endometriosis Pelvic inflammatory disease Ovarian cyst Myoma Chronic pelvic pain Urinary system infection Menometrorrhagia Obstructive vaginal or uterine congenital anomalies Secondary dysmenorrhea A history of major abdominal or pelvic surgery in the last 3 months Hormonal treatment in the last 6 months.

Ages: 18 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 22 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2019-06-06 (Actual); Study Completion 2019-07-02 (Actual)

PRIMARY OUTCOMES:
The primer outcome of the study was to investigate the effects of abdominal massage and exercise on the level of pain | 6 month
  Visuale Analogue Scale will be used to measure pain level at 3 menstrual cycle. The change from baseline in Visual Analog Scale at 3 menstrual cycle will be measured in the studied groups
The other primer outcome of the study was to investigate the effects of abdominal massage and exercise duration of pain. | 6 month
  Dysmenorrhea Symptom List will be used to measure degree of dysmenorrhea symptoms at 3 menstrual cycle. The findings seen in the presence of dysmenorrhea in females during 3 menstrual cycle will be measured by decrease at severity of scores belong to Dysmenorrhea Symptom List.

SECONDARY OUTCOMES:
The seconder outcome of the study was to investigate the effects of abdominal massage and exercise amount of menstruel bleeding | 6 month
  Pictorial Blood Loss Evaluation Table will be used to measure the amount of menstrual bleeding. The amount of menstrual bleeding will be measured by change from baseline in the pictorial index score at 3 menstrual cycle

CONTACTS AND LOCATIONS:
Overall Officials: Meryem Kurek Eken, Study Director — Aydin Adnan Menderes University
Locations (1):
- Meryem Kurek Eken, Aydin, Turkey (Türkiye)

REFERENCES:
- [Derived] Ozturk N, Gercek Oter E, Kurek Eken M. The effect of abdominal massage and stretching exercise on pain and dysmenorrhea symptoms in female university students: A single-blind randomized-controlled clinical trial. Health Care Women Int. 2023 May;44(5):621-638. doi: 10.1080/07399332.2022.2061973. Epub 2022 Aug 18. PMID 35980872